CLINICAL TRIAL: NCT00262717
Title: A Randomised Comparator Study to Assess the Relative Efficacy of Genotypic Versus Virtual Phenotypic Resistance Tests in Treatment Experienced Patients With HIV Infection for Whom a Change in Therapy is Indicated
Brief Title: Can Resistance Enhance Selection of Treatment? (CREST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Abbott (Industry); Boehringer Ingelheim (Industry); GlaxoSmithKline (Industry); Bristol-Myers Squibb (Industry); Merck Sharp & Dohme LLC (Industry); Roche Pharma AG (Industry); Virco (Industry); Diagnostic Technology (Industry); Perkin Elmer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVRP9901; ACTR012605000781640
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HIV Infection
Keywords: HIV drug resistance testing; Treatment Experienced
MeSH Terms: conditions — HIV Infections

ARMS (2):
- Group A: subjects assign to receive a GENOTYPE (Experimental): randomised prior to the selection of their new cART regimen
  Interventions: Diagnostic Test: Blood test: genotype testing
- Group B: subjects assign to receive a VIRTUAL PHENOTYPE (Experimental): randomised prior to the selection of their new cART regimen
  Interventions: Diagnostic Test: Blood test: genotype testing

INTERVENTIONS:
Diagnostic Test: Blood test: genotype testing

SUMMARY:
To compare two commercially available platforms for assessment of HIV drug resistance to determine which provides superior virological results.

We hypothesise that one test will be significantly superior to the other.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients taking combination antiretroviral therapy, with plasma HIV RNA> 2000copies/mL, who were willing to change ARVs and who provided informed consent.

Exclusion Criteria:

* Patients who were ARV naïve, who were experiencing an acute illness or judged to be unable to comply with the protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2001-03-01 (Actual); Primary Completion 2006-01-30 (Actual); Study Completion 2006-07-31 (Actual)

PRIMARY OUTCOMES:
The comparison between randomly assigned study arms in the mean area under the curve plasma HIV RNA at 48 weeks. | at 48 weeks follow-up

SECONDARY OUTCOMES:
Proportion of patients with undetectable plasma HIV RNA, Changes in CD4+ cell count, use of resistance test result in selecting new ART regimen | at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sean Emery, PhD, Study Chair — The National Centre in HIV Epidemiology and Clinical Research at the University of New South Wales
Locations (19):
- Australia (19):
  - Interchange General Practice, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Sydney Sexual Health Clinic, Sydney, New South Wales
  - AIDS Research Initiative, Sydney, New South Wales
  - Albion Street Centre, Sydney, New South Wales
  - Holdsworth House General Practice, Sydney, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Taylor Square Private Clinic, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Livingston Road Sexual Health, Sydney, New South Wales
  - QLD Health - AIDS Medical Unit, Brisbane, Queensland
  - Cairns Base Hospital, Cairns, Queensland
  - Gold Coast Sexual Health Clinic, Miami, Queensland
  - Care and Prevention Programme, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - Melbourne Sexual Health Centre, Melbourne, Victoria
  - Prahran Market Clinic, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Royal Perth Hospital, Perth, Western Australia